CLINICAL TRIAL: NCT06279585
Title: Physical Therapy in Patients Undergoing Allogeneic Hematopoietic Stem Cell Transplantation With a Diagnosis of Chronic Graft-versus-host Disease: A Randomized Clinical Trial.
Brief Title: Physical Therapy in Patients Undergoing Allo-HSCT With cGVHD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Raquel Perez Aguilar, Principal Investigator, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ECA GVHD
Record Dates: First submitted 2024-01-28; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Graft-versus-host-disease; Graft Versus Host Disease, Chronic; Stem Cell Transplant Complications; Hematological Malignancy; Hematologic Cancer
Keywords: Hematopoietic Stem Cell Transplantation; Graft versus host disease; Physiotherapy; Rehabilitation; Physical therapy; Exercise
MeSH Terms: conditions — Graft vs Host Disease; Bronchiolitis Obliterans Syndrome; Hematologic Neoplasms; Motor Activity | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants from both groups will undergo the three assessments and receive standard medical care.The patients in the experimental group will participate, at Time T1 (week 1 to 12), in a 12-week physiotherapy treatment program consisting of a total of 38 sessions: 2 health education sessions, 24 supervised combined exercise sessions, and 12 self-administered complementary exercise sessions.
  Interventions: Other: Physical therapy
- Control group (No Intervention): Participants from both groups will undergo the three assessments and receive standard medical care.
  The Control Group (GC), externally to the trial itself, for ethical reasons, considering potential benefits without risks, and as a strategy for blinding the study itself, will carry out the physiotherapy treatment program following the final assessment of the study, becoming a hybrid program under the same protocol.

INTERVENTIONS:
Other: Physical therapy — Health education sessions and combined therapeutic exercise sessions, based on muscular strength training and cardiorespiratory endurance.
  Arms: Experimental group

SUMMARY:
Allogeneic Hematopoietic Stem Cell Transplantation (alloHSCT) represents the only curative option for many patients diagnosed with various hematologic neoplasms. Procedure-related morbidity and mortality pose challenges to long-term outcomes and quality of life, especially among patients who develop chronic graft-versus-host disease (cGVHD). There is a gap in healthcare that comprehensively addresses the specific needs of these patients. Physical therapy as an adjuvant treatment, through therapeutic exercise involving muscle strength and cardiorespiratory endurance, has shown positive influences on health markers and serves as a strong medical ally in similar profiles. Although these strategies could be reproducible and potentially beneficial for cGVHD patients, research has been limited to date, with the role of physical therapy possibly underutilized in this field. Justification: Unaddressed medical gap with no rigorously scientific responses specific to cGVHD. Objectives: This project aims to conduct the first randomized clinical trial from a physical therapy perspective as an adjuvant treatment for patients undergoing alloHSCT diagnosed with cGVHD.

DETAILED DESCRIPTION:
Design: Prospective controlled clinical trial.

Location: Virgen del Rocío University Hospital, Hematology Unit.

Statistical analysis plan:The data will be analyzed using SPSS v.26 software for Windows and Epidat 4.2. All statistical tests will be conducted considering a 95% confidence interval (p-value <0.05). To compare the score of the main outcome measure, quality of life (score range 0-200), between the experimental and control groups, the t-test or Mann-Whitney test will be employed (depending on the normality of the data). The comparison will be conducted at three time points (T0, T1, and T2). Furthermore, multivariate analysis will be performed using generalized equations of repeated measures to determine score changes between the groups. Since it is a Likert scale-based score, the Friedman test will be used to compare score changes, employing the Bonferroni test for pairwise comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic Graft-Versus-Host Disease (cGVHD) treated at Virgen del Rocío University Hospital will be invited to participate in the trial (n=108), under the following eligibility criteria: Inclusion criteria:
* Adult (18 years or older); Underwent allogeneic hematopoietic stem cell transplantation (alloHSCT) diagnosed with cGVHD; No medical contraindication for moderate or high-intensity exercise; Proficiency in the Spanish language; Have access to the internet.

Exclusion Criteria:

* Unable to perform initial or final physical assessments; Having serious pre-existing conditions before the oncological diagnosis or diseases that are not or poorly controlled; Not signing or delivering the informed consent on the indicated date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life | Week 1, Week 6, and Week 13
  MEASURE NAME: Functional Assessment of Cancer Therapy - Bone Marrow Transplantation (FACT-BMT); VERSION: 4; NUMBER OF ITEMS: 50; RESPONSE SCALE: 5 point Likert-type scale; SCORING:Manual scoring template, some items are reverse scored. Higher score represents better quality of life.
Chronic Graft-Versus-Host Disease (cGVHD) symptom burden | Week 1, Week 6, and Week 13
  Modified Lee Chronic Graft-Versus-Host Disease Symptom Scale (mLSS) for 7 days. This is an instrument with 7 domains (skin, eyes, mouth, lungs, nutrition, energy, and psychiatry) and a total of 28 items to assess. The response options for "Please inform us if any of the following problems have bothered you in the last 7 days" range from 0 to 4 (Not at all, A little, Moderately, Quite a bit, Extremely). A difference of 5 to 6 points (standard deviation) will be considered clinically significant. Subscales range from 0 to 100, with a higher score indicating worse symptoms.

SECONDARY OUTCOMES:
Muscular strength | Week 1, Week 6, and Week 13
  Sit-to- Stand test y Handrig strength test
Cardiorespiratory fitness | Week 1, Week 6, and Week 13
  2-min Walk Test
Functional status | Week 1, Week 6, and Week 13
  Human Activity Profile (HAP)
Distress | Week 1, Week 6, and Week 13
  Distress-Thermometer
Mood | Week 1, Week 6, and Week 13
  "Mood Assessment Scale" (MAS); Designed to assess transient mood states, both positive and negative, in any individual at any time, through 16 items divided into four scales (depression, anxiety, hostility, and joy), each defined by 4 items and evaluated using the Likert scale, with scores ranging from 0 to 10. The values for each category are calculated by the mean. All 16 statements have the same structure; they all begin with the phrase "I feel" and end with an adjective describing a mood state.
Anxiety | Week 1, Week 6, and Week 13
  Hospital Anxiety and Depression Scale (HADS) questionnaire; The "Hospital Anxiety and Depression Scale questionnaire" (HADS); a useful tool for identifying anxiety and depression states in cancer patients and applicable during clinical practice. The two categories consist of one subscale each, with seven items rated from 0 to 4 points, with higher scores (in the range of 0 to 21) indicating anxious and depressive states. Participants should respond considering how they felt and/or behaved during the last seven days.
Biological markers | Week 1, Week 6, and Week 13
  Cytokines (interleukins) and lymphocytic populations as part of routine analysis. Blood sample.
Responses to medical treatment | Week 1, Week 6, and Week 13
  NIH Criteria

CONTACTS AND LOCATIONS:
Overall Officials: José Antonio P Simón, PHD, Study Director — Chief of Hematology at Virgen del Rocío University Hospital.
Locations (1):
- University of Seville; Manuel Siurot Avenue, no number, Seville, Spain

IPD SHARING:
Plan to Share IPD: Yes
Study protocol for a randomized clinical trial.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: When the study concludes; estimating by the end of the year 2025
Access Criteria: Both the study protocol and results, as well as the statistical plan, will be published in journals registered in the Journal Citation Report